CLINICAL TRIAL: NCT06504199
Title: A Prospective, Open-Label, Single-Arm Study of Obinutuzumab, Zanubrutinib, and Lenalidomide Followed Short-Cycle Cytarabine in First-Line Treatment of Mantle Cell Lymphoma
Brief Title: Obinutuzumab, Zanubrutinib, and Lenalidomide Followed Short-Cycle of Obinutuzumab and Cytarabine in Newly Diagnosed Mantle Cell Lymphoma
Acronym: ZGR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024010
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-04

CONDITIONS: Mantle Cell Lymphoma
Keywords: newly diagnosed; Mantle Cell Lymphoma; ZGR; Short-Cycle Cytarabine
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — obinutuzumab; zanubrutinib; Lenalidomide; Cytarabine

STUDY DESIGN:
Intervention Model Description: reated with 6 cycles of ZGR followed by a short cycle (3 cycles) of cytarabine + Obinutuzumab induction therapy. The maintenance regimen was selected according to patient risk stratification. Zanubrutinib in combination with lenalidomide was used for maintenance treatment in non-high-risk patients; maintenance treatment with zanubrutinib in combination with lenalidomide was allowed in high-risk patients after recovery of hemogram 2 months after treatment with chimeric antigen receptor T cells (CAR-T), with lenalidomide maintained for 1 year and zanubrutinib maintained for 2 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZGR followed short cycle of Obinutuzumab and Cytarabine (Experimental): All patients were treated with ZGR regimen for 6 cycles after enrollment, followed by 3 cycles of Obinutuzumab and Cytarabine in 28-day cycles. Obinutuzumab: 1000 mg, intravenous drip, administered on d1, d8 and d15 of the first cycle, and administered on the first day of each cycle starting from the second cycle. Zanubrutinib: 160 mg, bid, continuous oral. Lenalidomide: 20 mg/d, qd, oral, d1-d21.Cytarabine: for young tolerable patients, the dose is 2 g/m2, q12h, intravenous drip, d1-2ND for elderly/intolerant patients, the dose is 500 mg/m2, q12h, intravenous drip, completed 2-3 hours, d1-3. The specific dose is determined by the investigator according to the actual situation of the patient. Zanubrutinib for 2 years combination with Lenalidomide for 1 year was used for maintenance treatment in non-high-risk patients and in high-risk patients after recovery of hemogram 2 months after CAR-T.
  Interventions: Drug: Obinutuzumab; Drug: Zanubrutinib; Drug: Lenalidomide; Drug: Cytarabine; Biological: CAR-T

INTERVENTIONS:
Drug: Obinutuzumab — No dose adjustment of Obinutuzumab is allowed.
Drug: Zanubrutinib — Zanubrutinib was allowed to be titrated to 80 mg bid or 80 mg qd
Drug: Lenalidomide — Lenalidomide was allowed to be titrated to 15 mg/day (induction phase) or 5 mg/day (maintenance phase).
Drug: Cytarabine — The specific dose is determined by the investigator according to the actual situation of the patient.
Biological: CAR-T — zanubrutinib in combination with lenalidomide was allowed for maintenance treatment in high-risk patients for 1 year and zanubrutinib for 2 years after recovery of hemogram 2 months after CAR-T. High-risk Patients with any of the following conditions: Mantle cell lymphoma International Prognostic Index (MIPI-c) high-risk, blastic/pleomorphic type, TP53 mutation/deletion, CDKN2A deletion, MYC amplification/translocation, or incomplete response at induction stage; Non-high-risk group: no high-risk features.

SUMMARY:
This study aims to preliminarily explore the efficacy and safety of the combination of Obinutuzumab and Zanubrutinib plus Lenalidomide (ZGR) followed by a short cycle of cytarabine and Obinutuzumab in the induction treatment of newly diagnosed mantle cell lymphoma (MCL) . The investigators propose ZGR followed by a short cycle of Obinutuzumab and cytarabine could be an effective first-line treatment for MCL.

DETAILED DESCRIPTION:
Based on the clinical need for first-line treatment of MCL, this study proposed to enroll 39 patients with MCL who have not previously received any systemic therapy for MCL. All patients were treated with ZGR regimen for 6 cycles after enrollment, followed by 3 cycles of Obinutuzumab + cytarabine in 28-day cycles. For non-high-risk patients, lenalidomide and Zanubrutinib were used for maintenance; high-risk patients continued Lenalidomide and Zanubrutinib for maintenance following CAR-T cell therapy for 1 year for Lenalidomide and 2 years for Zanubrutinib. The primary endpoint of CRR and secondary endpoints (including ORR, PFS, DoR, and OS) were followed and recorded to explore the efficacy and safety of ZGR followed by a short cycle of Obinutuzumab and cytarabine induction therapy in treatment-naive MCL.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years, male or female;
2. Patients with pathologically (histologically or cytologically) confirmed MCL and at least one measurable lesion by Lugano criteria;
3. No prior systemic therapy for MCL;
4. Eastern Cooperative Oncology Group (ECOG) score of 0-2 points;
5. Normal function of vital organs, i.e. meeting the following criteria:

   a) Blood routine examination must be in accordance with (no blood transfusion, no use of hematopoietic factors and no use of drugs for correction within 14 days): i. Absolute neutrophil count (ANC) ≥ 1 × 10＾9/L; ii. Platelet count (PLT) ≥ 75 × 10＾9/L; b) Chemistry panel must meet the following criteria: i. Total bilirubin (TBIL) ≤ 2.0 × upper limit of normal (ULN); ii. Glutamic pyruvic transaminase (ALT), glutamic oxaloacetic transaminase (AST) ≤ 2.0 × ULN iii. Creatinine clearance ≥ 30 mL/min (Cockcroft-Gault formula); c) Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%;
6. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to the start of study medication and are willing to use a medically recognized highly effective contraceptive method (e.g., intrauterine device, contraceptive pill, or condom) during the study and within 6 months after the last dose of study drug; male subjects with partners of childbearing potential should be surgically sterile or agree to use an effective method of contraception during the study and within 6 months after the last dose of study drug;
7. The subjects voluntarily participate in the study and sign the informed consent form. They have good compliance and cooperate in the follow-up.

Exclusion Criteria:

1. Known central nervous system disease such as brain or meninges, including central nervous system lymphoma.
2. Congestive heart failure, Class III or IV (New York Heart Association, NYHA);
3. Other primary malignancies within the last 3 years (except non-melanoma skin cancer, curatively treated localized prostate cancer, carcinoma in situ of the cervix, or squamous epithelial endothelial lesions on PAP smear)
4. Previous use of investigational drugs;
5. Any active systemic viral, bacterial, or fungal infection requiring antimicrobial therapy within 2 weeks prior to the first dose of study drug;
6. Use of immunosuppressive agents, excluding nasal sprays and inhaled corticosteroids or physiological doses of systemic steroids (i.e., no more than 20 mg/day prednisone or its equivalent) within 7 days prior to the first dose of study drug
7. Allergic reactions, anaphylactic reactions and adverse drug reactions

   1. Severe allergic reactions to other monoclonal antibodies;
   2. Allergy or intolerance to infusion;
   3. Patients with a history of serious allergy to the investigational drug or its preventive medication;
8. Physical examination and laboratory findings

   1. Patients with congenital or acquired immunodeficiency, such as active hepatitis B virus (HBV DNA ≥ 500 IU/mL), hepatitis C (hepatitis C antibody positive, and HCV-RNA higher than the lower limit of detection of the analytical method) or combined hepatitis B and C co-infection;
   2. Pregnant or lactating women; patients with fertility are unwilling or unable to take effective contraceptive measures;
   3. Known history of positive human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS);
9. Any condition that, in the opinion of the investigator, may jeopardize the subject or may render the subject unable to meet or perform the study requirements;
10. Other conditions that the investigator considers inappropriate for entry into this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | up to the end of 9 cycles of treatment(each cycle is 28 days)
  defined as the proportion of patients with complete response as assessed by response to induction therapy using the 2014 Lugano criteria.

SECONDARY OUTCOMES:
overall response rate (ORR) | up to the end of 9 cycles of treatment(each cycle is 28 days)
  defined as the proportion of patients with complete or partial response as assessed by response to induction therapy.
Minimal residual disease (MRD) negative rate of | up to the end of 9 cycles of treatment(each cycle is 28 days)
  defined as the proportion of patients with MRD negative (less than 10-4) in bone marrow by flow cytometry after induction therapy in newly diagnosed patients with bone marrow invasion.
Progress-free survival (PFS) | up to 5 years
  defined as the time from the start of treatment to disease progression or death due to any cause.
Duration of tumor remission (DoR) | up to 5 years
  defined as the time from the first treatment response (including complete response and partial response) to the last assessment of response.
Overall survival (OS) | up to 5 years
  defined as the time from enrollment to death for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (2):
- China (2):
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality
  - Institute of Hematology and Blood Diseases Hospital ,Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No